CLINICAL TRIAL: NCT01880788
Title: Evaluation of Genetic Variants in Patients With Type 1 Neovascularization (Sub-retinal Pigment Epithelium Neovascularization) Who Lack Typical Findings of Age Related Macular Degeneration (AMD) But Present With Findings More Consistent With Long-standing Central Serous Chorioretinopathy (CSC).
Brief Title: Genetic Analysis of Chronic Central Serous Chorioretinopathy Masquerading as Neovascular AMD
Status: Completed | Type: Observational
Sponsor: Sequenom, Inc. (Industry)
Collaborators: Vitreous -Retina- Macula Consultants of New York (Other)
Responsible Party: Principal Investigator, K. Bailey Freund, MD, Clinical Associate Professor at NYU School of Medicine, Vitreous -Retina- Macula Consultants of New York
Other Study IDs: SCMM-AMD-107
Record Dates: First submitted 2013-05-16; First posted 2013-06-19 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Age Related Macular Degeneration; Choroidal Neovascularization; Central Serous Chorioretinopathy
Keywords: Age Related Macular Degeneration; Choroidal Neovascularization; Central Serous Chorioretinopathy
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization; Central Serous Chorioretinopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buccal cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- CNV secondary to CSC
- CSC without CNV
- CNV secondary to advanced AMD

SUMMARY:
The study will be designed as a case control evaluation to compare the genetic profiles of three groups of patients categorized according to diagnosis.

Group 1 - CNV secondary to CSC Group 2 - CSC without CNV Group 3 - CNV secondary to advanced AMD.

DETAILED DESCRIPTION:
To determine if patients presenting with type 1 neovascularization believed to be secondary to CSC are genetically distinct from typical CSC patients without neovascularization or patients presenting with choroidal neovascularization (CNV) secondary to advanced AMD. Disease associated markers detecting variants in ARMS 2, Complement Factor H (CFH) Complement component 3 (C3), Complement component 2 (C2) , Factor B (FB), VEGFA or other genetic polymorphisms associated with CNV will be evaluated to determine if the CSC neovascular group is genetically distinct from the CSC group without neovascularization or the advanced AMD group.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian
* 30 years and older (CSC)
* 50 years and older (Advanced AMD)
* Genders Eligible for Study: Both
* Completed Consent form
* Diagnosis of choroidal neovascularization in at least one eye

Exclusion Criteria:

* Patient age less than 30 years (CSC).
* Patient age less than 50 years (AMD).
* Presence of retinal disease involving the photoreceptors and/or outer retinal layers other than AMD and CSC such as high myopia, retinal dystrophies, retinal vein occlusion, diabetic retinopathy and uveitis or similar outer retinal diseases which have been present prior to the age of 30.
* Opacities of the ocular media, limitations of pupillary dilation or other problems sufficient to preclude adequate fundus photography.
* Missing informed consent
* Previous sample donation under this protocol

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen for routine visits at the offices of Vitreous Retina Macula Consultants of New York.
  Enrollment will include 150 subjects: 50 will be selected based on diagnosis of CNV secondary to CSC 50 will be selected based on diagnosis of CSC without neovascularization and 50 selected based on diagnosis of CNV secondary to advanced AMD.
Sampling Method: Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2012-11; Primary Completion 2015-03 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Total genetic burden | Baseline assessment
  The identification of individual genetic markers or a quantitative measure of total genetic burden associated with CNV secondary to CSC vs. CSC vs. CNV secondary to advanced AMD as meaured by the commercially available RetnaGene AMD assay.

CONTACTS AND LOCATIONS:
Locations (1):
- Vitreous Retina Macula Consultants of New York, New York, New York, United States